CLINICAL TRIAL: NCT03176290
Title: Non-Invasive Assessment of Graft Fibrosis After Living Donor Liver Transplantation: Is There Still a Rolefor Liver Biopsy?
Brief Title: Non-Invasive Assessment of Graft Fibrosis After Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Clinical professor, Ain Shams University
Other Study IDs: Assessment of liver fibrosis
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fibro-α score = (1.35 (numeric constant) +AFP (IU ml-1) × 0.009584 + aspartate aminotransferase (AST)/alanine aminotransferase(ALT) × 0.243 - platelet count (×109 l-1) × 0.001624). — Radiological investigations included Abdominal Doppler ultrasound, Magnetic Resonance Elastography(within 3 months of liver biopsy) and fibroscan.
  Other Names: Radiological investigations

SUMMARY:
The aim of this study is to compare prospectively the ability of MRE and Transient Elastography in detection and staging of allograft fibrosis in comparison to Liver biopsy in patients who underwent Living Donor Liver Transplantation for complications related to HCV.

DETAILED DESCRIPTION:
The study included Patients transplanted for HCV related disease diagnosed by positive serum PCR (HCV RNA) and liver biopsy with elevated liver enzymes and/orhyperbilirubinemia with Normal Abdominal Doppler ultrasound and MRCP.Other aetiology for liver disease as indication for transplantation and other causes of post-transplant abnormal liver profile as Post transplant biliary stricture or vascular liver diseases (if unresolved) were excluded from the study. Patients with active CMV infection(proved by positive CMV PCR or positive inclusion bodies by histopathology) were also excluded. All patients were subjected toFull history taking and thorough clinical examination, Laboratory investigations including CBC, Liver profile tests, Albumin, Bilirubin (Total and Direct), ALP(Alkaline phosphatase), AST(Aspartate aminotransferase), ALT (Alanine aminotransferase), INR (International Normalization Ratio),HCV RNA quantitative,CMV PCR, AST/ platelet ratio, Alpha feto-protein and fibro alpha score

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients who are candidate for LDLT due to HCV related ESLD and meeting the transplantation criteria of the Ain Shams Center of Organ Transplantation (Child Pugh score ≥ 7and MELD score ≥15).

Exclusion Criteria:

* Adult recipients who underwent LDLT due to other causes rather than HCV. Cardiopulmonary disease that cannot be corrected and is a prohibitive risk for surgery Acquired immunodeficiency syndrome (AIDS) Malignancy outside of the liver not meeting oncologic criteria for cure Hepatocellular carcinoma with metastatic spread Anatomic abnormalities that preclude liver transplantation Uncontrolled sepsis Acute liver failure with a sustained intracranial pressure >50 mmHg or a cerebral perfusion pressure <40 mmH Persistent non adherence with medical care and Lack of adequate social support Advanced age older than 65y.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent Living donor liver transplantation for HCV related disease
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
compare between liver biopsy and Magnetic Resonance Elastography (MRE) in assessment of liver fibrosis in HCV recipients after living donor liver transplantation | 6 months
  The aim of this study is to compare prospectively the ability of MRE and Transient Elastography in detection and staging of allograft fibrosis in comparison to Liver biopsy in patients who underwent Living Donor Liver Transplantation for complications related to HCV.

IPD SHARING:
Plan to Share IPD: Undecided